CLINICAL TRIAL: NCT00711893
Title: Feature Assessment Study for Indications Based Programming
Acronym: FASt-IBP
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Guidant Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: FASt-IBP 0408; feci 08/1644
Record Dates: First submitted 2008-07-07; First posted 2008-07-09 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Ventricular Tachycardia; Ventricular Flutter; Ventricular Fibrillation; Heart Failure
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Flutter; Ventricular Fibrillation; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICD and CRT-D: Patients indicated for an implantable defibrillator or cardiac resynchronization defibrillator
  Interventions: Device: Cognis 100-D, Teligen DR and VR 100 HE

INTERVENTIONS:
Device: Cognis 100-D, Teligen DR and VR 100 HE — Teligen is an implantable defibrillator for detection and termination of life threatening arrhythmias. Cognis includes in addition to these capabilities cardiac resynchronization therapy for patients having heart failure.

SUMMARY:
The purpose of this evaluation is to assess the acceptance level of specific programming recommendations based on the patient's clinical needs and primary indications when using the feature 'Indications Based Programming' (IBP) available in the ZOOMVIEW Software Application for the TELIGEN DR / VR and COGNIS family of devices compared to daily life programming chosen by physicians.

DETAILED DESCRIPTION:
"This study will focus on documenting the final parameter changes that are made in comparison to the IBP recommendations for a specific cardiovascular and arrhythmia history. It will therefore compare the device settings that were finally programmed during the last available follow up procedure to the last available parameter recommendations of IBP. IBP was designed to facilitate programming by providing customized parameter settings based on a patient's clinical needs and primary indication.

In order to further enhance the IBP feature for future device generations, additional data may be collected and evaluated on:

* Physician perception and satisfaction with the New User Interface (NUI) of the programming application;
* Motivation for adapting IBP recommendations for the final programming of the device;
* Device data that can be retrieved from patient data disks that may include but is not limited to, arrhythmia episode detail, pacing counter data; total and individual therapy data"

ELIGIBILITY:
Inclusion Criteria:

* indicated for implantation of an ICD or CRT-D device according local hospital implant criteria guidelines

  * Implanted or intended to be implanted with any CE-marked device approved for implant from the TELIGEN (single or dual chamber ICD) or COGNIS (CRT-D) family during first implant (no replacements)
  * Geographically stable patients who are available for follow-up at a study centre
  * Age 18 or above, or of legal age to give informed consent specific to national law

Exclusion Criteria:

Inability or refusal to sign the Patient Informed Consent

* Pregnant or planning to become pregnant
* Replacement device
* Enrolment in another clinical trial, study or evaluation
* Estimated life expectancy of less than six months per discretion of physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for the implant of an cardioverter defibrillator or cardiac resynchronization defibrillator defibrillator.
Sampling Method: Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2008-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients that are programmed by the physician to anything other than the recommended IBP setting | 6 Months

SECONDARY OUTCOMES:
- Degree of acceptance of IBP - Proportion parameters changed per patient - Differences between recommended and final programmed parameters - Total number of parameter changes from IBP recommendations - Frequency of changes made to a single parameter | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Goehl, MD, Principal Investigator — Klinikum Nuernberg
Locations (28):
- Austria (2):
  - KH der Elisabethinen Linz, Linz
  - KH der Barmherzigen Schwestern Ried/Innkreis, Ried
- Hartcentrum Hasselt - Dienst Cardiologie, Hasselt, Belgium
- Prince of Wales Hospital, Hong Kong, Hong Kong, China
- France (6):
  - EHRU de Brest - Hospital de la Cavale Blanche, Brest
  - CHU Dijon - Hospital du Bocage, Dijon
  - CHR Orléans - Hospital la Source, Orléans
  - CMC Parly II, Parly
  - CHU de St. Etienne-Hospital Nord, Saint-Priest-en-Jarez
  - CHU de Tours, Tours
- Germany (8):
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Praxis Dres. Bischoff/Lang, Erfurt
  - Klinikum Fulda, Fulda
  - Marienhospital Herne, Herne
  - Klinikum Kassel, Kassel
  - Praxis Schnabel der Praxisgemeinschaft Kardiologie Meissen, Meissen
  - Klinikum Nuernberg, Nuremberg
  - Klinikum Dorothea Christiane Erxleben Quedlinburg GmbH, Quedlinburg
- University Hospital of Heraklion, Heraklion, Greece
- Paul Stradina Clinical University Hospital, Riga, Latvia
- Netherlands (2):
  - Ziekenhius Rijnstate Arnhem, Arnhem
  - Amphia Ziekenhius Breda, Breda
- Narodny ustav srdcvych a cievnych chorob, Bratislava, Slovakia
- Spain (4):
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Son Llatzer, Palma de Mallorca
  - Clinico Universitario de Valladolid, Valladolid
  - Centro Miguel Servet, Zaragoza
- University Hospital of Geneva, Geneva, Switzerland